CLINICAL TRIAL: NCT04564937
Title: A Multicenter, Open-label, Multi-dose, Phase I / II Clinical Study to Evaluate Safety, Tolerability, Pharmacokinetics, Efficacy and Pharmacodynamic Characteristics of SCT510A in the Patients With Wet Age-related Macular Degeneration.
Brief Title: The Study of Drug SCT510A in Patients With Wet Age-related Macular Degeneration (wAMD)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SCT510A-A101
Record Dates: First submitted 2020-09-16; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Wet Age-related Macular Degeneration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SCT510A dose level 1 treatment (Experimental): SCT510A(0.625mg), Vitreous injection, injection once every 4 weeks，three times continuously
  Interventions: Drug: SCT510A
- SCT510A dose level 2 treatment (Experimental): SCT510A(1.25mg), Vitreous injection, injection once every 4 weeks，three times continuously
  Interventions: Drug: SCT510A
- SCT510A dose level 3 treatment (Experimental): SCT510A(2.0mg), Vitreous injection, injection once every 4 weeks，three times continuously
  Interventions: Drug: SCT510A
- SCT510A dose level 4 treatment (Experimental): SCT510A(2.5mg), Vitreous injection, injection once every 4 weeks，three times continuously
  Interventions: Drug: SCT510A

INTERVENTIONS:
Drug: SCT510A — SCT510A of 0.625mg、1.25mg、2.0mg、2.5mg,IVT

SUMMARY:
Multicenter ，open-label, multi-dose study to evaluate the safety and tolerability in patients with wAMD treated with intravitreal recombinant humanized anti-VEGF monoclonal antibody（SCT510A）

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form;
2. Age≥45 years，≤80 years，male or femal;
3. The study eye must meet the following criteria： Diagnosis of wAMD； Primary or recurrent active subfoveal or parafoveal choroidal neovascularization (CNV) lesions secondary to AMD； Total area of all types of lesions ≤12 optic disc areas（30mm2）； Best-corrected visual acuity of the study eye 70 letters or worse(Snellen equivalent of 20/40 or worse)； No optometric media opacity and pupil shrinkage.
4. Best-corrected visual acuity of the fellow eye 19 letters or better（Snellen equivalent of 20/400 or better）.

Exclusion Criteria:

1. The study eye suffers structural damage of retinal which involves fovea，and the investigator assess that there is a risk of retinal detachment；
2. Significant afferent pupillary defect (APD) in the study eye；
3. The study eye has no lens( except intraocular lens) or posterior capsular rupture of the lens；
4. In addition to AMD，there are other obvious eye diseases/conditions，such as pseudoexfoliation syndrome，rhegmatogenous retinal detachment，macular hole，diabetic retinopathy and diabetic macular disease which need to be treated；
5. CNV caused by other causes other than wAMD, such as vascular stripe disease, ocular histoplasmosis, case myopia, trauma, etc；
6. Uncontrolled glaucoma in the study eye (defined as IOP≥25mmHg after antiglaucoma treatment),or recevied glaucoma filtering surgery；
7. History of vitreous hemorrhage in the study eye within 2 months before the first administration；
8. Active inflammation or infection in either eye, such as conjunctivitis,keratitis, scleritis, endophthalmitis, or uveitis，ect；
9. Previous intraocular surgery ，or laser therapy for wAMD(as photodynamic therapy,transpupillary thermotherapy,etc.) in the study eye within 3 months before the first administration；
10. Previous intraocular or periocular injection of anti-VEGF or corticosteroid drugs (such as ranibizumab, bevacizumab, conbercept, aflibercept, brolucizumab, pegaptanib sodium, anecortave acetate, triamcinolone acetonide, etc.) in either eye within 3 months before the first administration；
11. History of allergy to fluorescein sodium or indocyanine green；
12. PLT≤100×109/L；thrombin time and prothrombin time exceed the upper limit of normal range (based on the laboratory normal value of clinical trial institution), and the abnormality is clinically significant according to the evaluation of the investigators；
13. Abnormal liver and kidney function；
14. Uncontrolled blood pressure control，systolic blood pressure≥160mmhg ,or diastolic blood pressure≥100mmhg；
15. History of surgery within one month before the first administration, or current non-healing wound, ulcer, or fracture，etc；
16. Patients with any of the following serious systemic diseases，such as serious mental, neurological, cardiovascular, respiratory and other system diseases and malignant tumors, systemic immune system diseases, diabetes mellitus with uncontrolled blood sugar(HbA1c>10%), disseminated intravascular coagulation and significant bleeding tendency；
17. Suffering from systemic infectious diseases requiring oral, intramuscular or intravenous administration；
18. Pregnant, lactating women and the patients who can not take contraceptive measures.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-11-06 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting toxicity(DLT) | From Day 0 up to Day 14
  Incidence of dose-limiting toxicities up to the Day 14 visit
Maximum tolerated dose(MTD） | From Day 0 up to Day 140
  Maximum tolerated dose

SECONDARY OUTCOMES:
PK profile | From Day 0 up to 84 days
  Change of SCT510A drug concentration in the blood with time
Cmax | From Day 0 up to 84 days
  The maximum blood concentration after SCT510A drug enters the bloodstream
Tmax | From Day 0 up to 84 days
  Time to the Maximum Concentration of SCT510A
t1/2 | From Day 0 up to 84 days
  Elimination Phase Half-life of SVT510A
Biomarker | From Day 0 up to 84 days
  Detection of free VEGF concentration
Immunogenicity | From Day 0 up to 112 days
  Positive rate of ADA and NAb
central retina thickness（CRT） | From Day 0 up to 140 days
  Changes in CRT compared to the baseline
Macular edema volume | From Day 0 up to 140 days
  Changes in Macular edema volume compared to the baseline
Best corrected visual acuity（BCVA） | From Day 0 up to 140 days
  Changes in BCVA compared to the baseline